CLINICAL TRIAL: NCT02640287
Title: Expression of Ku70/XRCC6 and Others NHEJ Components in Waldenström's Macroglobulinemia in Comparison With Others B-cell Lymphoproliferative Disorders and Normal B Cells.
Brief Title: Expression of Ku70/XRCC6 in Waldenström's Macroglobulinemia
Acronym: WAL-KU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Aurore PERROT, Principal Investigator, Central Hospital, Nancy, France
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2015-A01516-43
Record Dates: First submitted 2015-12-22; First posted 2015-12-28 (Estimated); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Waldenström Macroglobulinemia
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Waldenström macroglobulinemia (Experimental): Patients with diagnosis of Waldenström macroglobulinemia
  Interventions: Biological: Blood or bone marrow samples
- Others B-cell malignancies (Experimental): Patients with diagnosis of Chronic Lymphocytic Leukemia, Splenic Marginal Zone Lymphoma or Multiple Myeloma
  Interventions: Biological: Blood or bone marrow samples
- Healthy subjects (Other): Control healthy subjects without B-cell malignancy
  Interventions: Biological: Blood or bone marrow samples

INTERVENTIONS:
Biological: Blood or bone marrow samples

SUMMARY:
Waldenström's macroglobulinemia is a rare disease whose pathophysiology remains at present poorly understood, although a recurrent mutation (L265P MYD88) has recently been described. Unlike other lymphoproliferative disorders, there is a defect in isotype switching, mechanism involving AID and NHEJ complex. Using a two-dimensional electrophoresis technology, our group showed that MW had a specific proteomic profile, and one of the differentially expressed proteins is Ku70 (encoded by XRCC6 belonging to NHEJ complex) .

The investigators purpose to explore the mechanisms of underexpression of Ku70/XRCC6 (genetic or epigenetic modification) in comparison with other lymphoid malignancies and normal B cells.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years, affiliated to the social regimen
* Written consent collected

MW group :

* Patient with a diagnosis of MW according to WHO criteria (based on the results of serum protein electrophoresis, bone marrow analysis with immunophenotyping, cytogenetic analysis and mutation L265P MyD88)

Other SLP :

* Patient with diagnosis of Chronic Lymphocytic Leukemia, Splenic Marginal Zone Lymphoma or Multiple Myeloma

Healthy volunteers :

* volunteers without blood disorders

Exclusion Criteria:

* Women of childbearing age who do not have an effective means of contraception
* Pregnant or nursing
* Demonstration of a kappa or lambda monotype on B lymphocytes
* healthy volunteer with B-cell malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2016-02; Primary Completion 2020-06-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Measure of ratio Ku70/XRCC6 | Baseline
  Comparing the average level of expression of Ku70 in B cells measured in patients of WM, in patients other SLP and in healthy subjects (without MW and other SLP) , matched for age ( +/- 5 years) and sex

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Nancy, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No